CLINICAL TRIAL: NCT06039722
Title: Prospective, Multicenter, Single-arm Clinical Trial Evaluating the Safety and Efficacy of the Pulse Field Ablation System in Combination With the Pulse Field Ablation Catheter for the Treatment of Paroxysmal Atrial Fibrillation.
Brief Title: Safety-and-effectiveness Clinical Evaluation of Nanosecond-pulse Ablation for Atrial Fibrillation
Acronym: SCENA-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Pulsecare Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMTCT2022001
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2023-09

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Pulse Field Ablation Catheter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): Each subject underwent pulse ablation catheter ablation
  Interventions: Device: Pulse ablation catheter

INTERVENTIONS:
Device: Pulse ablation catheter — Pulse ablation catheter is used to ablate the junction of left atrium and pulmonary vein, removing pulmonary vein potential

SUMMARY:
This study is expected to include 166 subjects and Conducted at 11 research centers；The expected 12 month treatment success rate of using research instruments is 65%.

Principle evaluation indexes：

1. Immediate success rate of surgery Immediately success of the surgery: complete pulmonary vein electrical isolation was achieved after ablation.
2. Immediate success rate of surgery=number of patients with immediate success of surgery/number of cases in subjects × 100%
3. Treatment success rate at 12 months after surgery Treatment success: Between 3 months and 12 months after ablation, there were no episodes of atrial fibrillation/atrial flutter/atrial tachycardia (duration ≥ 30 seconds, with clear electrocardiogram confirmation) without the use of antiarrhythmic drugs.

Treatment success rate=number of successful cases of postoperative treatment in subjects/number of cases in subjects × 100%

Secondary evaluation indexes：

1. The occurrence of hospitalization or emergency treatment due to symptoms caused by atrial arrhythmias during follow-up at 6 and 12 months after surgery;
2. Device performance evaluation;

Safety evaluation indexes：

1. The occurrence of death, stroke, or transient ischemic attack;
2. The occurrence of surgical related complications, such as vascular puncture complications (pseudoaneurysm, arteriovenous fistula, etc.), heart perforation, atrial esophageal fistula, phrenic nerve injury, pulmonary vein stenosis (symptomatic), etc;
3. Clinically significant vital signs and related examinations;
4. The occurrence of other adverse events and serious adverse events during the trial period.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following conditions to be enrolled:

1. 18 to 80 years of age, gender is not limited
2. Patients with a clinical diagnosis of paroxysmal atrial fibrillation confirmed by ECG
3. Patients who were to undergo catheter ablation of atrial fibrillation
4. Those who agreed to participate in this study and voluntarily signed the informed consent form

Exclusion Criteria:

Subjects were excluded if they met one of the following conditions:

1. Patients who have had ablation for atrial fibrillation
2. Patients with left ventricular ejection fraction (LVEF) <35%.
3. Patients with an anteroposterior diameter of the left atrium (echocardiography) >50 mm
4. Preoperative detection of a definite thrombus in the left atrium
5. Patients with cardiac function class (NYHA) III-IV
6. Patients with second-degree (type II) or third-degree atrioventricular block
7. Patients with significant congenital heart defects (including atrial septal defect, ventricular septal defect, arterial ductus arteriosus, transposition ofthe grea, or severe pulmonicvalve, but not including foramen ovale persistens)
8. Patients with implanted prosthetic valves or the presence of severe heart valve disease, who are not suitable for ablation for atrial fibrillation
9. Patients with artificial cardiac pacemaker or implantable cardioverter defibrillator (ICDs)
10. Patients diagnosed with hypertrophic obstructive cardiomyopathy, chronic obstructive pulmonary disease, or myxoma
11. Patients who need to undergo left atrial appendage closure in the same surgery
12. Patients found to have atrial flutter preoperatively and judged unsuitable by the investigators, or patients with atrial parasystolic tachycardia (non-pulmonary venous origin) or paroxysmal supraventricular tachycardia
13. Patients with active systemic infection who are judged unsuitable for interventional therapy by the investigators
14. Patients with systemic bleeding tendencies that preclude surgery or patients with renal failure undergoing hemodialysis
15. Patients who have had a myocardial infarction or any interventional/open heart surgery (except coronary angiography) within 3 months
16. Patients who have had a stroke (except asymptomatic stroke) or transient ischemic attack within 3 months
17. Patients with significant contraindications to interventional procedures or with an expected survival of <1 year who are judged by the investigator to be incapable of undergoing ablative procedures
18. Females who are pregnant or breastfeeding or who are planning to have children during the study period
19. Patients who have participated in a clinical trial of another drug or medical device within 3 months
20. Patients who, in the opinion of the investigator, are not suitable for participation in this clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Immediate success rate of surgery | After surgery 20 minutes later
  Immediate success rate of surgery Immediately success of the surgery: complete pulmonary vein electrical isolation was achieved after ablation.
  Immediate success rate of surgery Immediately success of the surgery: complete pulmonary vein electrical isolation was achieved after ablation.
  Immediate success rate of surgery Immediately success of the surgery: complete pulmonary vein electrical isolation was achieved after ablation.
  Immediate success rate of surgery=number of patients with immediate success of surgery/number of cases in subjects × 100%
Treatment success rate | Between 3 months and 12 months after ablation
  Treatment success rate at 12 months after surgery Treatment success: Between 3 months and 12 months after ablation, there were no episodes of atrial fibrillation/atrial flutter/atrial tachycardia (duration ≥ 30 seconds, with clear electrocardiogram confirmation) without the use of antiarrhythmic drugs.
  Treatment success rate=number of successful cases of postoperative treatment in subjects/number of cases in subjects × 100%

SECONDARY OUTCOMES:
numer of cases of the the occurrence of hospitalization or emergency treatment | Between 0 months and 12 months after ablation
  The occurrence of hospitalization or emergency treatment due to symptoms caused by atrial arrhythmias during follow-up at 6 and 12 months after surgery;
Device performance evaluation | surgery period
  Device defects of the clinical trial equipment

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Sun Yat-sen University （Sun Yat-sen Memorial Hospital）, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie S, Lai H, Jia F, Zhang Z, Wang Y, Yin Y, Chen Q, Huang H, Liu Q, He J, Yang P, Wang J. High-Repetition-Frequency Nanosecond Pulsed Field Ablation for Paroxysmal Atrial Fibrillation: 12-Month Outcomes From the SCENA-AF Trial. Circ Arrhythm Electrophysiol. 2026 Feb 4:e014236. doi: 10.1161/CIRCEP.125.014236. Online ahead of print. PMID 41636062